CLINICAL TRIAL: NCT06608186
Title: Can Drospirenone be Used to Prevent LH Surge in Controlled Ovarian Stimulation in PCOS Cases
Brief Title: Can Drospirenone be Used to Prevent LH Surge in Controlled Ovarian Stimulation in PCOS?!
Acronym: PPOS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ahmed Saad (Other)
Responsible Party: Sponsor-Investigator, Ahmed Saad, Professor of Obsterics & Gynecology, Benha University
Organization: Benha University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hawaa-10
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: PCOS (Polycystic Ovary Syndrome)
Keywords: PCOS; PPOS; Drospirenone; Gn antagonist
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — cetrorelix; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Intervention Model Description: 50 case in this novel trial. 25 in each group will be randomized after taking 5 days of ovarian stimulation to either drospirenone tablet/d or cetrorelix injection/d till the day of hCG.
Who Masked: Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drospirenone (Experimental): 25 cases will receive drospirenone in the form of 1 tablet / d from day 5 of stimulation till hCG trigger day
  Interventions: Drug: Drospirenone drug
- cetrorelix (Active Comparator): 25 cases will receive cetrorelix from day 5 of stimualtion till hCG trigger day
  Interventions: Drug: Cetrorelix drug

INTERVENTIONS:
Drug: Cetrorelix drug — a drug injection daily sc. from day 5 of stimulation till hCG trigger day
  Other Names: cetrorelix
  Arms: cetrorelix
Drug: Drospirenone drug — A drug drospirenone in the form of 1 tablet / d from day 5 of stimulation till hCG trigger day
  Arms: Drospirenone

SUMMARY:
The goal of this clinical trial is to learn if drospirenone can work to prevent LH surge in controlled ovarian stimulation in PCOS cases undergoing ART cycles. The main questions it aims to answer are:

Can drospirenone prevent LH surge in controlled ovarian stimulation in PCOS cases ? Can it prevent the occurance of ovarian hyperstimulation?

Researchers will compare drospirenone to cetrorelix (A well known drug for such cases) to see if drospirenone works the same way.

Participants will:

Take drospirenone or cetrorelix from stimulation day 5 ( 5 days of ovarian stimulation) till day of hCG trigger

- monitoring will be done before the cycle and through the cycles with vaginal ultrasound assessment and lab testing

DETAILED DESCRIPTION:
The goal of this novel clinical trial is to study if drospirenone can work to prevent LH surge in controlled ovarian stimulation in PCOS cases undergoing ART cycles in comparison to a gold standard drug cetrorelix:

All PCOS cases: 50 case in this novel trial. 25 in each group will be randomized after taking 5 days of ovarian stimulation to either drospirenone tablet/d or cetrorelix injection/d till the day of hCG.

At the day of hCG, lab testing will be done in addition to ultrasound assessment by transvaginal probe. the tests are: progesterone, E2, LH.

Assesment will be done for the number quality of follicles and the number quality of embryos developed, development of OHSS, vitrification/thawing of embryos after 1 month then the clinical and chemical pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* PCOS was diagnosed according to the Rotterdam consensus criteria (two out of three of the following criteria):

  1. oligo- or anovulation
  2. clinical and/or biochemical signs of hyperandrogenism
  3. polycystic ovaries).
* A diagnosis of congenital adrenal hyperplasia, Cushing's syndrome, androgen-producing tumours, hyperprolactinemia and thyroid dysfunction were all rulled out.

Exclusion Criteria:

* age 38 years
* basal FSH level 12 mIU/mL
* previous ovarian surgery
* congenital uterine anomaly anomaly, intrauterine adhesion and male partner with non-obstructive azoospermia.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female gender phenotypically and genetically
Enrollment: 50 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-19 (Actual); Study Completion 2025-01-19 (Actual)

PRIMARY OUTCOMES:
number of cases to develop OHSS | 1 week
  cases that will develop OHSS
number of embryos | 5 days
  number of embryos developed

SECONDARY OUTCOMES:
clinical pregnancy rate | 15 days after embryo transfer
  serum pregnancy test after thawing of the embryos and embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed s saad, phD, Study Director — Professor of OB & GYN
Locations (1):
- Hawaa Fertility center, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the protocol excel sheet
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months
Access Criteria: 6 months